CLINICAL TRIAL: NCT03749473
Title: Evaluation of the Novel Use of Gamification With Alternative Goal-setting Experiences
Acronym: ENGAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Mitesh Patel, Assistant Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 831258
Record Dates: First submitted 2018-11-14; First posted 2018-11-21 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Atherosclerotic Cardiovascular Disease
Keywords: Physical Activity; Goal-Setting; Gamification
MeSH Terms: conditions — Atherosclerosis; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (Active Comparator): Participants receive a daily message with their step count on the prior day to serve as an active control for 24 weeks (daily performance feedback). No other interventions during the 24-week study
  Interventions: Behavioral: Daily performance feedback
- Choice + Immediate (Experimental): Participants choose a step goal between 1000-3000 steps greater than their baseline (choice). They are asked to reach their full step goal upon intervention start (immediate). They will be in a gamification intervention for the first 16 weeks and then receive only daily feedback during the 8-week follow-up
  Interventions: Behavioral: Choice + Immediate; Behavioral: Daily performance feedback; Behavioral: Gamification
- Choice + Gradual (Experimental): Participants are asked to choose a step goal between 1000-3000 steps greater than their baseline (choice). They will be asked to increase their step goal by even increments of 12.5% each week for the 8 weeks of the ramp-up period (gradual). After the 8-week ramp-up period, they will be asked to maintain the step goal for the study. They may change their goal within the range at anytime. They will be in a gamification intervention for the first 16 weeks and then receive only daily feedback during the 8-week follow-up
  Interventions: Behavioral: Choice + Gradual; Behavioral: Daily performance feedback; Behavioral: Gamification
- Assigned + Immediate (Experimental): Participants in this arm will be assigned a step goal 2000 steps greater than their baseline (assigned). They will be asked to reach their full step goal as soon as the intervention begins (immediate). They will be in a gamification intervention for the first 16 weeks and then receive only daily feedback during the 8-week follow-up
  Interventions: Behavioral: Assigned + Immediate; Behavioral: Daily performance feedback; Behavioral: Gamification
- Assigned + Gradual (Experimental): Participants in this arm will be assigned a step goal 2000 steps greater than their baseline (assigned). They will be asked to achieve their step goal of 2000 steps incrementally over the 8 weeks of the ramp-up period (gradual). After the first 8 weeks, they will be asked to maintain their full step goal of 2000 for the the study. They will be in a gamification intervention for the first 16 weeks and then receive only daily feedback during the 8-week follow-up
  Interventions: Behavioral: Assigned + Gradual; Behavioral: Daily performance feedback; Behavioral: Gamification

INTERVENTIONS:
Behavioral: Choice + Immediate — Participants in the choice + immediate goal arm will choose a step goal and must attempt to achieve this new step goal immediately at the start of the study.
  Arms: Choice + Immediate
Behavioral: Choice + Gradual — Participants in the choice + gradual goal arm will choose a step goal and will gradually work towards the chosen step goal over the first 8-weeks of the study.
  Arms: Choice + Gradual
Behavioral: Assigned + Immediate — Participants in the assigned + immediate goal arm will be assigned a step goal and must attempt to achieve this new step goal immediately at the start of the study.
  Arms: Assigned + Immediate
Behavioral: Assigned + Gradual — Participants in the assigned + gradual goal arm will be assigned a step goal and will gradually work towards the chosen step goal over the first 8-weeks of the study.
  Arms: Assigned + Gradual
Behavioral: Daily performance feedback — Participants will receive daily performance feedback on their daily step count.
Behavioral: Gamification — All participants in the intervention arms will be entered into a gamification platform that has points and levels designed to incorporate insights from behavioral economics.
  Arms: Assigned + Gradual; Assigned + Immediate; Choice + Gradual; Choice + Immediate

SUMMARY:
To use a randomized controlled trial to test the effectiveness of four goal-setting strategies within a gamification intervention to increase physical activity among adults at elevated risk for ASCVD.

DETAILED DESCRIPTION:
Atherosclerotic cardiovascular disease (ASCVD) is the leading cause of mortality in the United States. While increased physical activity can reduce this risk, less than half of adults in the United States meet the minimum recommendation guidelines for physical activity. Gamification, or the application of game design elements to non-game settings, has demonstrated promise in increasing physical activity when designed using insights from behavioral economics. However, the best way to design goal-setting within these interventions has not been well-examined. In this randomized controlled trial, the investigators will evaluate the effectiveness of four different goal-setting strategies within a gamification intervention to increase physical activity among adults with elevated risk for ASCVD. The trial will include a 2-week run-in period to estimate a baseline, followed by an 8-week introductory phase, an 8-week maintenance phase, and then after the intervention is completed an 8-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older;
* ability to read and provide informed consent to participate in the study;
* diagnosis of clinical ASCVD or a 10-year ASCVD risk score ≥ 7.5% calculated according to the 2013 ACC/AHA guidelines;
* Smartphone or tablet compatible with application for the wearable activity tracking device.

Exclusion Criteria:

* Conditions that would make participation infeasible such as inability to provide informed consent, illiteracy or inability to speak, read, and write English;
* conditions that would make participation unsafe such as pregnancy or being told by a physician not to exercise;
* already enrolled in another study targeting physical activity;
* any other medical conditions or reasons he or she is unable to participate in a physical activity study for 24 weeks;
* baseline step count of 10,000 steps or greater.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change in mean daily steps from baseline to maintenance period. | Baseline to weeks 9-16
  The primary outcome is change in mean daily steps from baseline to weeks 9-16 (maintenance period).

SECONDARY OUTCOMES:
Change in mean daily steps from baseline to follow-up period. | Baseline to the weeks 17 to 24
  The secondary outcome is change in mean daily steps from baseline to the weeks 17 to 24 (follow-up period).

OTHER OUTCOMES:
Change in minutes of MVPA from baseline to maintenance and follow-up periods. | Baseline to weeks 9-16 and weeks 17-24
  An exploratory outcome is change in minutes of moderate-to-vigorous physical activity (MVPA) from baseline to weeks 9-16 (maintenance) and weeks 17-24 (follow-up period).
Change in minutes of sleep from baseline to maintenance and follow-up periods. | Baseline to weeks 9-16 and weeks 17-24
  An exploratory outcome is change in minutes of sleep from baseline to weeks 9-16 (maintenance) and weeks 17-24 (follow-up period).

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh S Patel, MD, MBA, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available

REFERENCES:
- [Derived] Patel MS, Bachireddy C, Small DS, Harrison JD, Harrington TO, Oon AL, Rareshide CAL, Snider CK, Volpp KG. Effect of Goal-Setting Approaches Within a Gamification Intervention to Increase Physical Activity Among Economically Disadvantaged Adults at Elevated Risk for Major Adverse Cardiovascular Events: The ENGAGE Randomized Clinical Trial. JAMA Cardiol. 2021 Dec 1;6(12):1387-1396. doi: 10.1001/jamacardio.2021.3176. PMID 34468691